CLINICAL TRIAL: NCT04151550
Title: Evaluation of the Safety and Efficacy of the Laser Scleral Microporation Procedure to Restore Visual Function and Range of Accommodation
Brief Title: Safety & Efficacy of the Laser Scleral Microporation Procedure (Philippines)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ACE Vision Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVG-PHIL-2019-02
Record Dates: First submitted 2019-11-01; First posted 2019-11-05 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Presbyopia
Keywords: Presbyopia; Sclera; Laser Scleral Microporation
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- AVG LSM Procedure (Other): Ace Vision Group LSM procedure performed on both eyes.
  Interventions: Device: Bilateral Laser Scleral Microporation procedure

INTERVENTIONS:
Device: Bilateral Laser Scleral Microporation procedure — Device: Laser Scleral Microporation
  Partial depth scleral microporations with an Er:YAG laser in a predetermined pattern.

SUMMARY:
A minimally invasive procedure for treating presbyopia is being evaluated to determine if there is improvement in near and intermediate vision after treatment.

DETAILED DESCRIPTION:
This is a prospective, controlled, single-center clinical study to evaluate the safety and efficacy of the Laser Scleral Microporation Procedure.

Laser Scleral Microporation Procedure is a treatment to restore visual and accommodative function in presbyopic patients. The subjects are bilaterally treated with the Laser Scleral Microporation procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to understand and sign an informed consent;
2. Willing and able to attend postoperative examinations per protocol schedule;
3. 48 years of age or greater, of either gender or any race;
4. Less than (<) 1.00D of astigmatism in each eye, measured by manifest refraction;
5. Mean Refractive Spherical Equivalent (MRSE) of less than or equal to 0.50D for distance vision;
6. Uncorrected Distance Visual Acuity (UDVA) is better than or equal to 20/40 (logMAR 0.30) in each eye, and a Corrected Distance Visual Acuity (CDVA) is better than or equal to 20/25 (logMAR 0.10) in each eye;
7. Demonstrate stereopsis of 100 seconds of arc or better using a Stereo Fly test with near correction;
8. In good ocular health with the exception of presbyopia;
9. Presbyopia as demonstrated by:

   1. Currently wearing reading glasses and/or bifocals with an ADD of +1.50D or more at 40cm in each eye; and
   2. Reduced near visual acuity at 40cm when corrected for distance (DCNVA) of 20/50 (logMAR 0.40) or worse in each eye;
10. Intraocular pressure (IOP) ≥ 11mmHg and ≤ 30 mmHg in each eye without IOP-lowering medication;
11. Less than or equal to (≤) 0.50D difference between the manifest refraction spherical equivalent and the cycloplegic refraction spherical equivalent;
12. If the subject has had Laser Vision Correction (LVC) within 1-2 years prior to the LSM procedure, stable distance refraction is present, defined as ≤ 0.50D variation of refraction in the 12 months prior to the LSM procedure. Manifest refraction spherical equivalent (MRSE) cannot vary more than 0.50D from current spectacles that are at least 12 months of age, or from a documented refraction at least 12 months prior to the preoperative baseline exam; if baseline data is available.
13. Completed a washout period of two weeks (14 days) prior to LSM procedure from prior treatment with:

    a) With prior medical clearance: non-steroidal anti-inflammatory drugs (NSAIDs), blood thinners, aspiring and other substances which may increase bleeding; b) Anti-oxidants, which could affect blood thinning: (i) Any antioxidant supplements (e.g., Vitamin E, Acai, Ocuvite, greater than 1000mg of Omega-3, etc.); (ii) Antioxidant food supplements, such as shitake mushroom, mushroom extract and oral antioxidants

Exclusion Criteria:

1. Self-reported current pregnancy or breast-feeding, or plans to become pregnant during the entire study period;
2. History of ocular trauma or prior ocular surgery, or expected to require retinal laser treatment or other ocular surgical intervention;
3. Presence of ocular pathology other than cataract such as:

   1. Amblyopia or strabismus
   2. Corneal abnormalities or disease
   3. History of Dry Eye treatments/devices
   4. Pupil abnormalities (e.g., corectopia, Adie's)
   5. Capsule or zonular abnormalities
   6. Intraocular inflammation
   7. Retinal/macular disease or pathology
   8. Glaucoma (any type)
4. History of prior ocular surgery, including:

   1. Previous corneal surgery (e.g., penetrating keratoplasty, DSEAK/DSEK/DMEK, lamellar keratoplasty), except for LASIK, SMILE, EpiLASEK, or PRK;
   2. Previous anterior or posterior chamber surgery (e.g., vitrectomy, laser iridotomy) with the exception of uncomplicated phacoemulsification with intraocular lens implantation;
   3. Previous retinal surgery (e.g, retinal break, repair related to ocular trama or detachment, or pathology that is likely to require surgical intervention such as lattice degeneration.
5. Known pathology that may affect visual acuity and/or are predicted to cause future acuity losses to a level of 20/30 (logMAR 0.18) or worse (e.g., macular degeneration);
6. Keratoconus or keratoconus suspect with CDVA of less than (<) 20/20 (logMAR 0.00) at distance;
7. Near visual acuity at 40cm equivalent to their distance vision with distance correction (i.e., no evident effect of reduced accommodative range);
8. Use of systemic or ocular medications that may affect vision (the use of any miotic or cycloplegic agent is specifically contraindicated);
9. Acute or chronic disease or illness that could increase the operative risk or confound the study outcome(s) (e.g., diabetes mellitus, immunocompromised, connective tissue disease);
10. Uncontrolled systemic or ocular disease;
11. Any abnormality preventing reliable applanation tonometry in EITHER eye;
12. Undilatable pupil such that one cannot examine the periphery of the retina;
13. Functional eye preference, defined as phoria measuring over 15 prism diopters (PD) horizontally and/or over 2 PD vertically, any strabismus, or suppression.
14. History of scleral ectasia, scleritis, or episcleritis: or thin sclera < 400 microns, as determined by taking the average of three measurements with ultrasound biomicroscopy (UBM) pachymetry or ocular coherence tomography;
15. History of nuclear sclerosis LOCS III grade 2 or worse and/or other cataracts reducing CDVA or OSI > 2.5;
16. Known allergies to study medications including topical steroids, antibiotics and NSAIDs;
17. Per Principal Investigator (PI) discretion

Min Age: 48 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Binocular Distance Corrected Near Visual Acuity (DCNVA) @40cm | 12 months postoperative
  Binocular DCNVA is measured with ETDRS charts placed in 40cm distance. This assessment is performed under photopic lighting conditions.

SECONDARY OUTCOMES:
Autorefraction | 1 week; 1 month; 3 months; 6 months; 12 months; 18 months & 24 months postoperative
  An autorefractor or automated refractor is a computer-controlled machine used during an eye examination to provide an objective measurement of a subject's refractive error.
Monocular Uncorrected Distance Visual Acuity (UDVA) @4m | 1 day; 1 week; 1 month; 3 months; 6 months; 12 months; 18 months & 24 months postoperative
  UDVA is measured with ETDRS charts placed at 4m distance. This assessment is performed monocularly under photopic lighting conditions.
Binocular Uncorrected Distance Visual Acuity (UDVA) @4m | 1 week; 1 month ; 3 months; 6 months; 12 months; 18 months & 24 months postoperative
  UNVA is measured with ETDRS charts placed at 4m distance. This assessment is performed binocularly under photopic lighting conditions.
Monocular & Binocular Uncorrected Intermediate Visual Acuity (UIVA) @60cm | 1 week 1 month; 3 months 6 months; 12 months; 18 months & 24 months postoperative
  UIVA is measured with ETDRS charts placed at 60cm distance. This assessment is performed monocularly, then binocularly under photopic lighting conditions.
Monocular & Binocular Uncorrected Near Visual Acuity (UNVA) @40cm | 1 week; 1 month; 3 months; 6 months; 12 months; 18 months & 24 months postoperative
  UNVA is measured with ETDRS charts placed at 40cm distance. This assessment is performed monocularly, then binocularly under photopic lighting conditions.
Manifest Refraction | 1 week; 1 month; 3 months; 6 months; 12 months; 18 months & 24 months postoperative
  This is the manual way to determine the best lenses, by placing various lenses in front of the subject's eyes and asking questions. The manifested refraction is measured by means of a phoropter and ETDRS charts at 4m. The data contains values for sphere, cylinder and axis of cylinder. This data will also be used to calculate the Manifest Refractive Spherical Equivalent (MRSE). This assessment is performed under photopic lighting conditions
Monocular & Binocular Best Corrected Distance Visual Acuity (CDVA) @4m | 1 week; 1 month; 3 months; 6 months; 12 months; 18 months & 24 months postoperative
  CDVA is measured with ETDRS charts placed at 4m distance using best aided corrective glasses. This assessment is performed monocularly, then binocularly under photopic lighting conditions.
Monocular & Binocular Distance Corrected Intermediate Visual Acuity (DCIVA) @60cm | 1 week; 1 month; 3 months; 6 months; 12 months; 18 months & 24 months postoperative
  DCIVA is measured with ETDRS charts placed at 60cm distance using corrective glasses for far distance. This assessment is performed monocularly, then binocularly under photopic lighting conditions.
Monocular Distance Corrected Near Visual Acuity (DCNVA) @40cm | 1 week postoperative; 1 month postoperative; 3 months postoperative; 6 months postoperative; 12 months postoperative; 18 months postoperative, 24 months postoperative
  Monocular DCNVA is measured with ETDRS charts placed in 40cm distance using corrective glasses for far distance. This assessment is performed monocularly under photopic lighting conditions.
Monocular Best Corrected Near Visual Acuity (DCNVA) @40cm | 1 week postoperative; 1 month postoperative; 3 months postoperative; 6 months postoperative; 12 months postoperative; 18 months postoperative, 24 months postoperative
  Monocular CNVA is measured with ETDRS charts placed in 40cm distance using corrective glasses for near distance (reading prescription). This assessment is performed monocularly under photopic lighting conditions.
Accommodative Amplitude using binocular & monocular minus lens to blur | 1 week; 1 month; 3 months; 6 months; 12 months; 18 months & 24 months postoperative
  The amplitude of accommodation is the maximum potential increase in optical power that an eye can achieve in adjusting its focus. The amplitude of accommodation will be assessed binocularly first at distance with an introduction of minus power over the distance prescription to stimulate accommodation. Instruct the subject to focus on 20/20 line of the ETDRS charts at 4m, and slowly add minus power in -0.25D steps until the subject reports first sustained blur on the line. Record the dioptric value where the subject reports the first sustained blur. Subtract the distance prescription from this value to obtain the Accommodative Amplitude using this method repeat three times). This assessment is performed binocularly first, then monocularly under photopic lighting conditions.
IReST | 1 week; 1 month; 3 months; 6 months; 12 months; 18 months & 24 months postoperative
  The International Reading Speed Texts (IReST) consists of paragraphs of text (approx. 130 words per text) which is a standardized assessment of reading speed. The reading speed will be measured using the IReST using the subject's reading prescription determined at each visit. This assessment will be performed under photopic lighting conditions.
Stereoacuity | 1 week; 1 month; 3 months; 6 months; 12 months; 18 months & 24 months postoperative
  Stereopsis, or depth perception, is based on the horizontal retinal image disparity between the two eyes. Stereoacuity, which is a threshold measure of the acuteness of this depth perception, provides an indication of the level of sensory binocularity an subject has. Stereoacuity will be measured using a the Precision Vision Stereo Fly test at 40cm with the subject's reading prescription. For this test, the reading prescription determined at each visit will be used and the assessment will be performed under photopic lighting conditions.
Contrast Sensitivity | 1 month postoperative; 12 months postoperative; 24 months postoperative
  Contrast sensitivity is the subject's ability to distinguish the foreground from the background.
  This will be measured using ETDRS (Sloan Revised Low Contrast Chart 2425) optotypes with 10% contrast while wearing distance correct placed in 4m distance. For this assessment will be performed under photopic lighting conditions.
Wavefront Aberrometry | 1 week; 1 month; 3 months; 6 months; 12 months; 18 months & 24 months postoperative
  The iTrace (Tracey Technologies, Houston, TX) measures aberrometry at distance 60cm and 40cm. Measurements will be performed uncorrected and corrected using the distance correction in loose lenses held in the Tracey trial frames. Higher order on lower order aberrations will be recorded using distance correction at distance, 60cm and 40cm.
Effective Range of Focus | 1 week; 1 month; 3 months; 6 months; 12 months & 24 months postoperative
  The iTrace (version 5.3.1 or higher, Tracey Technologies, Houston, TX) wavefront aberrometer is used for the DOF testing. The iTrace measures aberrometry at distance using the distance prescription in a trial frame, as well as at 60cm and 40cm using a near rod. Objective measures will be performed to assess the change in EROF based upon the location of the visual target.
Optical Scatter | 1 week; 1 month; 3 months; 6 months; 12 months & 24 months postoperative
  The HD Analyzer determines the Objective Scattering Index (OSI) which determines how a point source of light is imaged on the retina (recommended version 2400 -Keeler, Malver, PA).
Intraocular Pressure | 1, Day, 1 week; 1 month; 3 months; 6 months; 12 months; 18 months & 24 months postoperative
  Intraocular Pressure will be measured using Goldmann applanation tonometry. Tow measurements will be performed per eye at each visit. If there is more than 2mmHg between the two readings, a third reading will be performed. The value will be an average.
UBM Accommodation | 1 month; 12 month & 24 month postoperative
  An ultrasound eye exam that makes a more detailed image. The VuMAX HD (Sonomed Escalon, NY) is the recommended device for evaluation .

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Jackson, MD, Study Director — Ace Vision Group
Locations (1):
- Asian Eye Institute, Makati City, Philippines

IPD SHARING:
Plan to Share IPD: No